CLINICAL TRIAL: NCT02360267
Title: Pediatric Bipolar Registry
Acronym: PBR
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jair Soares, Professor, Principal Investigator, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-12-0673
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Bipolar Disorder; Depression; Mania; Psychosis
Keywords: Bipolar Disorder; Pediatric; Offspring; Depression; Mania; Children of parents who suffer from Bipolar disorder
MeSH Terms: conditions — Bipolar Disorder; Depression; Mania; Psychotic Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of the Pediatric Bipolar Registry (PBR) is to provide a comprehensive assessment regarding the diagnosis and treatment of pediatric bipolar disorder to children and adolescents with any current mood state and/or children/adolescents who are offspring of a parent with bipolar disorder (BD) type I or II and their families.

DETAILED DESCRIPTION:
Data collected will be utilized to perform a retrospective chart review to include measure outcomes and de-identified demographic information detailed in the attached case report forms. In each case where a diagnosis of bipolar disorder I, bipolar disorder II, or bipolar disorder NOS is determined, the child/adolescent will be added to the PBR and provided with information about local providers that are qualified to treat their diagnosis. Each subject can elect to be notified about future research studies s/he may qualify for. Furthermore, the investigators will provide ongoing newsletters with useful information that addresses the latest research underway in the field with the families. If requested, the investigators will provide a written report to their current provider detailing our evaluation. The potential for a breach in confidentiality always exists; however, information that is obtained will be stored in password a protected database and locked file drawers in locked offices; data will have identifying information sheered from it to prevent loss of confidentiality, and all staff must sign confidentiality certificates. If child abuse is detected, the research team is obligated to follow mandatory state reporting laws. To the investigators' knowledge, there is no registry for Pediatric Bipolar Disorder in the city of Houston or the state of Texas that provides the comprehensive evaluation that we are proposing for these children and adolescents and their families. Therefore, this will be a novel service within this division that will provide research to families and potential clients for providers managing these families across the State of Texas.

ELIGIBILITY:
Inclusion Criteria

1. Age 6-17 years old at time of initial visit.
2. Any current mood state Diagnosis of a DSM- IV Bipolar Disorder, Type I, Type II and NOS.
3. Offsprings of a parent diagnosed with Bipolar Disorder Type I or Type II.

Exclusion Criteria

1. Pervasive Developmental Disorder (PDD) (and/or PDD NOS)
2. Mental Retardation/Intellectual Disability
3. Severe Neurological Disorder that affects cognitive status (e.g., epilepsy, traumatic brain injury, tubular sclerosis).
4. Schizophrenia
5. Uncontrolled or severe medical problem

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children ages 6-17 who may suffer from Bipolar Disorder (BP I, BP II, or BP-NOS) or whose parents suffer from Bipolar Disorder (BP I or BP II).
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2013-08-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Course of diagnosis (per MINI kid interview) | 1 year
  AIM I:
  The goal of the Pediatric Bipolar Registry (PBR) is to provide a comprehensive assessment regarding the diagnosis of pediatric bipolar disorder to children and adolescents with any current mood state and/or children/adolescents who are offspring of a parent with bipolar disorder (BD) type I or II. Data collected will be utilized to perform a retrospective chart review to include measure outcomes and de-identified demographic information detailed in the attached case report forms. Each of these steps will allow result in a comprehensive Pediatric Bipolar Registry database.

SECONDARY OUTCOMES:
Changes in Young Mania Rating Scale (YMRS) and Childhood Depression Rating Scale (CDRS) scores | 2 years
  AIM II:
  In each case where a diagnosis of bipolar disorder I, bipolar disorder II, or bipolar disorder NOS is determined, the child/adolescent will be added to the Pediatric Bipolar Registry (PBR) and provided with information about local providers that are qualified to treat their diagnosis. Each subject can elect to be notified about future research studies s/he may qualify for. Furthermore, we will provide ongoing newsletters with useful information that addresses the latest research underway in the field with the families. If requested, we will provide a written report to their current provider detailing our evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Jair C Soares, MD, Principal Investigator — UT Health Science Center at Houston
Locations (1):
- UT Center of Excellence on Mood Disorders, Houston, Texas, United States